CLINICAL TRIAL: NCT02668471
Title: Ultrasound-guided Compared With Traditional Palpation Radial Artery Cannulation in Critically Ill Children
Brief Title: U/S Guided vs. Traditional Palpation for Radial Artery Cannulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Nattachai Anantasit, Principle investigator, Pediatric Department, Ramathibodi Hospital, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ID-09-58-14
Record Dates: First submitted 2016-01-22; First posted 2016-01-29 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultrasound guided (Experimental): Radial artery catheters will be placed with the assistance of bedside ultrasound.
  Interventions: Procedure: Ultrasound
- traditional method (Active Comparator): Radial artery catheters will be placed by the palpation technique only.
  Interventions: Procedure: traditional method

INTERVENTIONS:
Procedure: Ultrasound — ultrasound at radial site and measure the size and depth of radial artery and perform radial artery cannulation
  Arms: Ultrasound guided
Procedure: traditional method — Radial artery catheters will be placed by the palpation technique only.
  Arms: traditional method

SUMMARY:
The purpose of this study is to compare the efficacy of ultrasound- guided with the traditional palpation radial artery cannulation in critically ill children.

DETAILED DESCRIPTION:
Arterial catheterization is often performed in critically ill patients for continuous hemodynamic monitoring and blood sampling. However, insertion of radial artery catheter with traditional palpation may be technically challenging, particularly in pediatric patients. There are few published studies on the use of ultrasound guidance for radial-artery catheter placement and mostly they were elective surgery children which received inhalation or deep sedative medication. Recently no setting published in pediatric intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients who required radial artery cannulation for hemodynamic monitoring or frequent blood samples in intensive care unit

Exclusion Criteria:

* Wound at area of cannulation
* Can not palpate or weak radial artery pulse

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08-30 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
first attempt success rate of radial artery catheter insertion | 5 minute

SECONDARY OUTCOMES:
time to success of radial artery catheter insertion | 15 minute

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatric,Ramathibodi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huang HP, Zhao WJ, Wen F, Li XY. Application of ultrasound-guided radial artery cannulation in paediatric patients: A systematic review and meta-analysis. Aust Crit Care. 2021 Jul;34(4):388-394. doi: 10.1016/j.aucc.2020.09.001. Epub 2020 Oct 21. PMID 33097369